CLINICAL TRIAL: NCT03143296
Title: The Effects of Reverberation on Speech Understanding in MED-EL Cochlear Implant Recipients
Brief Title: Reverberation Effects on MED-EL Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Med-El Corporation (Industry)
Responsible Party: Principal Investigator, Sandra Prentiss, Associate Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20170198
Record Dates: First submitted 2017-04-26; First posted 2017-05-08 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current recipient of a Med-El cochlear implant (Experimental): Participants who have received a MED-EL cochlear implant as a standard of care for treatment of hearing loss. Participants are tested at one time point with a simulated reverberant environment.
  Interventions: Other: Simulated reverberant environment
- Future Med-El Recipient (Active Comparator): Cochlear implant candidates not yet implanted and chose Med-El device as standard of care for treatment of hearing loss. Participants are tested at 3 time points over 6 months in a simulated reverberant environment.
  Interventions: Other: Simulated reverberant environment

INTERVENTIONS:
Other: Simulated reverberant environment — Reverberant environments simulate real-life situations mimicking a living room, classroom and auditorium. Each simulation lasts up to 2 hours.

SUMMARY:
The purpose of this study is to investigate speech understanding in simulated reverberant environments with MED-EL cochlear implant recipients.

DETAILED DESCRIPTION:
The study will determine if electrode length and coding strategy effect performance. The investigator will also study performance over time with new recipients.

ELIGIBILITY:
Inclusion Criteria:

* MED-EL current cochlear implant recipients of the Flex 24 or 28 will be included
* Minimum of 6 months experience with their cochlear implant
* Minimum of 10 new adult Med-El recipients of the Flex 24 or Flex 28 electrodes
* Patient at the University of Miami

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Speech Performance | Up to six months
  Speech performance recorded as percent correct compared to different electrode lengths.
Coding strategy | Two hours
  Speech scores, in percent correct, recorded from simulated reverberant speech tests will be compared between fine structure and envelope coding strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Prentiss, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Department of Otolaryngology, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No